CLINICAL TRIAL: NCT02419014
Title: Cranial Electrotherapy for Military Beneficiaries With Restless Legs Syndrome
Acronym: CES in RLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 52H13
Record Dates: First submitted 2015-04-02; First posted 2015-04-17 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Restless Legs Syndrome
Keywords: cranial electrotherapy; cranial electrical stimulation; restless legs syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Participants in this group will continue receiving their previously prescribed therapy during the 8 week data collection period.
- Active CES Device (Active Comparator): The Alpha-Stim® device is a Class II FDA-approved device for the delivery of cranial electrotherapy using microcurrents that are delivered via two electrodes worn on the earlobes. Active CES devices will be pre-programmed by the manufacturer to deliver a bipolar, asymmetric rectangular waveform at a current of 100 µa, a level that is generally undetectable by the wearer of the device. At these settings, the manufacturer recommends a treatment duration of 60 minutes. Participants will not be able to alter the settings in any way.
  Interventions: Device: Active CES Device Alpha-Stim®
- Sham CES Device (Placebo Comparator): The inactive (sham) devices look identical to the active device but are inactivated by the manufacturer so as not to deliver any electrical current.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Active CES Device Alpha-Stim® — The Alpha-Stim® device is a Class II FDA-approved device for the delivery of cranial electrotherapy using microcurrents that are delivered via two electrodes worn on the earlobes. Active CES devices will be pre-programmed by the manufacturer to deliver a bipolar, asymmetric rectangular waveform at a current of 100 µa, a level that is generally undetectable by the wearer of the device. At these settings, the manufacturer recommends a treatment duration of 60 minutes. Participants will not be able to alter the settings in any way.
  Other Names: Alpha-Stim®; Cranial electrotherapy stimulator; Cranial electical stimulation therapy; microcurrent electrical therapy
  Arms: Active CES Device
Device: Sham Device — The inactive (sham) devices look identical to the active device but are inactivated by the manufacturer so as not to deliver any electrical current.
  Arms: Sham CES Device

SUMMARY:
The purpose of this study is to assess the feasibility and effectiveness of Cranial Electrical Stimulation (CES) therapy in treating symptoms of Restless Legs Syndrome (RLS). Participants will be randomly assigned to one of three groups, a usual care (control group), an active CES device group and a sham (inactive) CES device group. Those who are enrolled in one of the device groups will not know which type of device they have (blinding). Those enrolled in the usual care group and sham groups will ultimately have the option to use the active device after they complete the study. Study length for participants is 8 weeks.

DETAILED DESCRIPTION:
Restless Legs Syndrome (RLS) is a chronic neurologic disease that causes painful and distressing dysesthesias in the lower extremities at night affecting sleep quality and greatly influencing general overall health. Leading theories as to the cause of RLS symptoms point to a deficiency of central nervous system dopamine levels. Cranial Electrical Stimulation (CES) is a therapy that has been shown to affect activity in dopaminergic regions of the brain. The purpose of this study is to assess the feasibility and efficacy of CES therapy in the management of symptoms of RLS. The overall study design will use mixed methods. The specific aims for the experimental analysis are to (1) determine the feasibility of the implementation of a CES treatment regimen in a population of military beneficiaries with RLS by monitoring levels of interest in the study, recruitment time, attrition rates, and adherence to the study protocol; and (2) gather preliminary data using CES to compare differences in RLS symptom severity and quality of life in individuals randomized to one of three study groups: a usual care group, an inactive (sham) device group, or an active CES device group. Because the personal impact of living with RLS has not been explored fully in the published literature, a third aim is (3) to describe the experience of individuals coping with the chronic symptoms of RLS and the impact of this disorder on their quality of life. Measurements of RLS symptom severity and quality of life will be collected over a period of 8 weeks and group differences over time will be analyzed using mixed linear models. Qualitative interview data will be analyzed using descriptive phenomenological methods. Findings from this study will inform the design and implementation of a larger study to establish the effectiveness of CES on RLS symptoms. Qualitative findings will provide much needed information on the priorities for future research and clinical management based on patients' perspectives. The ultimate goal of the research is to identify and to evaluate the comparative effectiveness of non-pharmacological treatments for RLS symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Department of Defense Health Care Beneficiary
* A diagnosis of RLS, using criteria established by the International Restless Legs Study Group
* Currently symptomatic
* A period of 4 weeks of stable medication usage
* Over the age of 18
* Able to read, write and understand English.

Exclusion Criteria:

* Pacemaker or other implanted electrical device
* Pregnancy or breastfeeding
* Inadequately treated primary cause of RLS (i.e., iron deficiency) based on screening laboratory testing
* Lack of a formal diagnosis of RLS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in International Restless Legs Syndrome Study Group Rating Scale (IRLS) from baseline and weekly for 8 weeks post intervention | At baseline then every week for 8 weeks
  The IRLS consists of 10 questions, each with 5 possible responses geared towards assessing severity that range from no symptoms (0 points) to very severe symptoms (4 points). Scoring: Points for each response are added together to create a possible range of 0-40 with higher scores indicating worsening severity. Reliability and Validity: The IRLS demonstrated high internal consistency on 2 separate testing sessions (Cronbach's α of 0.93 and 0.95, respectively). Test/retest reliability demonstrated a correlation coefficient of 0.87 and paired t-test demonstrated stability over time.

SECONDARY OUTCOMES:
Qualitative Data Interview | Approximately 30-60 minute interview at any point during the study enrollment
  The purpose of this interview is to learn more about the lived-experience of RLS from those suffering from it in an effort to direct future research and treatment priorities
Change in The Hopkins Restless Legs Syndrome Quality of Life Scale (RLS-QOL) from baseline at 4 and 8 weeks post intervention | At baseline then at weeks 4 and 8
  The RLS-QOL consists of 18 total items measuring the domains of life impact, employment/work and sexual interest. Scoring: 10 of the items are added together to represent overall life impact, 6 items address employment/work and 2 address sexual interest. Higher scores are indicative of a higher quality of life. Reliability and Validity: The RLS-QOL demonstrated high internal consistency on 2 separate testing periods (Cronbach's α of 0.82 and 0.87, respectively). Validity was assessed by comparison to the IRLS (moderate correlation -0.68 and -0.67). The instrument was further assessed for sensitivity to change by demonstrating a significant difference (p < 0.0001) in the overall life impact score after treatment.
Change in the RAND 36-item Health Survey (RAND-36) from baseline at 4 and 8 weeks post intervention | At baseline then at weeks 4 and 8
  The scale consists of 36 items incorporating 8 domains of health: physical functioning; role limitations related to physical health; role limitations related to emotional health; energy/fatigue; emotional well-being; social functioning; pain; and general health. Scoring: A scoring key accompanies the instrument that links the specific item numbers to domains and instructs the scorer through conversion from the raw score to a scale score. Higher scores indicate higher quality of life. Reliability and Validity: Internal consistency of all domains was assessed with Cronbach's α ranging from 0.78 to 0.93, indicating high reliability.
Change in the Fatigue Severity Scale (FSS) from baseline weekly for 8 weeks post intervention | At baseline then every week for 8 weeks
  The FSS consists of 9 items for which participants identify their degree of agreement with the item on a 7-point Likert scale. Scoring: The FSS is scored by adding the numbers that are circled by participants and dividing by 9 to obtain an average score, which ranges from 1-7. Reliability and Validity: The FSS demonstrated high internal consistency in reliability testing with an overall Cronbach's α of 0.88. Test/retest stability over time demonstrated a correlation coefficient of 0.84. In t-tests assessing for responsiveness to change over time, clinical improvement after treatment for fatigue was associated with significant decreases in FSS score (p < 0.01).
Change in the Pittsburgh Sleep Quality Index (PSQI) from baseline at 4 and 8 weeks post intervention | At baseline then at weeks 4 and 8
  The PSQI (58) consists of 19 self-rated questions intended to discriminate between good sleepers and poor sleepers by measuring sleep habits on 7 different sleep domains: (1) subjective sleep quality; (2) sleep latency; (3) sleep duration; (4) habitual sleep efficiency; (5) sleep disturbances; (6) use of sleep medications; and (7) daytime dysfunction. Scoring: Scores are organized into the seven domains, which added together yield one global score ranging from 0-21 points. A lower score indicates low difficulty and a higher score indicates more severe difficulty within the identified domains. The seven domains combined have an overall reliability of 0.83 indicating high internal validity.

CONTACTS AND LOCATIONS:
Overall Officials: Terri L Yost, PhD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Tripler Army Medical Center, Honolulu, Hawaii, United States